CLINICAL TRIAL: NCT03543306
Title: An Open-label, Multicenter, Phase II Study of Dabrafenib and Trametinib in Patients With Non-small Cell Lung Cancer Harboring V600E BRAF Mutation
Brief Title: Dabrafenib and Trametinib in Patients With Non-small Cell Lung Cancer Harboring V600E BRAF Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-We Kim, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARTER_BRAF
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Lung Cancer Metastatic; BRAF V600E
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: daborafenib plus trametinib — Dabrafenib 150 mg twice daily and trametinib 2 mg once daily

SUMMARY:
This is a Phase II, non-randomized, open-label study to assess the efficacy, safety, and tolerability of dabrafenib and trametinib in stage IV disease to subjects with BRAF V600E mutant advanced non-small cell lung cancer. Subjects will receive dabrafenib 150 mg bid and trametinib 2 mg once daily in combination therapy and continue on treatment until disease progression, death, or unacceptable adverse event.

ELIGIBILITY:
Inclusion Criteria:

Subjects with histologically or cytologically confirmed, unresectable stage IIIB/IV NSCLC that carries a V600 BRAF mutation, as per NGS ECOG performance status of 0 to 2 Male or female; ≥ 18 Subjects with measurable lesion (using RECIST 1.1 criteria) Subjects must have archival tissue sample available, collected either at the time of diagnosis of NSCLC or any time since Patients who have progressed during or after 1st line or 2nd line therapy prior to the first dose of dabrafenib/trametinib. For patient who have received prior platinum containing adjuvant, neoadjuvant, or definitive chemoradiation for locally advanced disease, those treatments are regarded as 1st line if the progression has occurred < 12 months from last therapy.

Subjects who meet the following criteria:

Absolute neutrophil count (ANC) >1.5 x 109/L Platelet count >100 x 109/L Serum creatinine >1.5 x upper limit of normal (ULN) AST (SGOT) and ALT (SGPT) > 3 x upper limit of normal (ULN) (If there is Liver Metastasis > 5 x upper limit of normal (ULN)) Total bilirubin>1.5 x upper limit of normal (ULN) the progression has occurred < 12 months from last therapy. Patients with asymptomatic brain metastasis could be eligible. Provision of written informed consent prior to any study specific procedures

Exclusion Criteria:

Any major operation or irradiation within 4 weeks of baseline disease assessment Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms Subjects with chemotherapy naïve or those who already had received two lines of chemotherapy including immunotherapy or targeted therapy.

Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or cervical cancer in situ.

Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome, 2° or more AV Block and uncontrolled hypertension) Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of drug pneumonitis, hypersensitivity pneumonitis, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).

Pregnant or lactating female Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with IPs for the duration of participation:

Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm) Strong inhibitors or strong inducers of CYP2C8 and CYP3A4 Unstable or increasing doses of corticosteroids enzyme-inducing anticonvulsive agents herbal supplements Patients who have received thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  ORR is a proportion of patients with a best overall response defined as complete response or partial response by RECIST1.1

SECONDARY OUTCOMES:
Duration of response | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  DOR is calculated as the time from the date of the first document of complete remission (CR) or partial remission (PR) to the first documented preogressive disease (PD) or death due to any cause for patients with PR or CR.
Progression-free survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  . PFS is defined as time from the first dose of investigational products (IPs) to progression or death due to any cause. OS is defined as time from the first dose of IPs to death due to any cause.
Overall survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
Disease control rate | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  DCR is calculated as the proportion of patients with best response of CR, PR and SD.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided